CLINICAL TRIAL: NCT03025984
Title: Adherence to a Diabetes Care Regimen Following Text Message Intervention in Pregnant Women With Diabetes
Brief Title: Texting for Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Dorothea Mostello, MD, Principal Investigator, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22596
Record Dates: First submitted 2017-01-11; First posted 2017-01-20 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
Keywords: diabetes pregnancy text message
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Texting (Active Comparator): Patients in the "Texting" group will receive reminders based on their individual disease treatment. A text message shall be sent one day (12 to 36 hours) before appointments to remind about the appointment and with instructions to bring glucose and food records to the appointment. If medication changes are made at the appointment, the patient will receive a text message reminder the day after her appointment to reinforce the regimen. Postpartum patients who had GDM will receive a text message reminder to complete their glucose tolerance test. A reminder will be sent at 2 weeks postpartum followed by a reminder at 6 weeks and 10 weeks postpartum if the testing is not completed.
  Interventions: Behavioral: Texting
- No texting (No Intervention): Patients in the contact control group will be enrolled in the text4baby program with assistance from a healthcare provider. As the study will conclude upon the patient's postpartum visit, she will be offered the option of discontinuing messages, which otherwise would continue through the infant's first year of life.

INTERVENTIONS:
Behavioral: Texting — patient adherence to her recommended care regimen after intervention of a text message reminder and education system
  Arms: Texting

SUMMARY:
Diabetes is a common complication of pregnancy that increases risks for both the mother and baby. Poorly controlled diabetes has been associated with very large babies, congenital heart defects, stillbirth, birth trauma, and maternal infections among other complications. Patients with diabetes in pregnancy require more frequent prenatal visits and fetal evaluation, and must shoulder the burden of mastering management of a complicated care regimen. With the ever-expanding world of technology, more healthcare practices are using cell phones, texting, and social media to interact with patients. Use of this technology has been successful in management of chronic diseases and as reminder systems. The investigators propose a randomized clinical trial to investigate patient adherence to recommended care regimen after intervention of a text message reminder and education system.

DETAILED DESCRIPTION:
As a part of routine care, pregnant women without known diabetes undergo screening and testing for gestational diabetes either with a two-hour glucose tolerance testing or a one-hour glucose challenge test followed by a three-hour glucose tolerance test in the event of failure of the one-hour test.

Women who have been given the diagnosis of gestational diabetes mellitus (GDM) by failing this diabetes testing and who meet the inclusion and exclusion criteria shall be approached and offered enrollment in the study. Women with known type 2 diabetes mellitus (T2DM) (pre-gestational diabetes) and women diagnosed elsewhere with GDM who meet the inclusion and exclusion criteria will be offered enrollment when they establish prenatal care. Patients who consent to participate in the study shall be randomized to either the intervention or the contact control group. For randomization purposes, an equal number of notecards will be made for the two groups. These will all be placed in sealed envelopes and shuffled. At the time of patient inclusion, an envelope will be selected by the consenting practitioner. If a patient declines receiving text messages but consents to have her medical record reviewed for adherence to her diabetes care regimen and glycemic control, she will be enrolled in the standard of care control group. A baseline hemoglobin A1c (HbA1c) is obtained.

Patients in all groups shall receive initial diabetes education and started on an individualized diabetic diet regimen. Patients with GDM who develop a requirement for either oral medication or insulin will remain in the same group to which they were initially randomized. An HbA1c level is obtained every one to three months during pregnancy as well as near the time of delivery.

Patients in the intervention group will receive reminders based on their individual disease treatment. A text message shall be sent one day (12 to 36 hours) before appointments to remind about the appointment and with instructions to bring glucose and food records to the appointment. If medication changes are made at the appointment, the patient will receive a text message reminder the day after her appointment to reinforce the regimen. Postpartum patients who had GDM will receive a text message reminder to complete their glucose tolerance test. A reminder will be sent at 2 weeks postpartum followed by a reminder at 6 weeks and 10 weeks postpartum if the testing is not completed. Women with T2DM will be reminded to bring glucose and food records to their postpartum visits. Participants will be contacted through Google Voice which is a Google system requiring a secure login and password.

Patients in the contact control group will be enrolled in the text4baby program with assistance from a healthcare provider. As the study will conclude upon the patient's postpartum visit, she will be offered the option of discontinuing messages, which otherwise would continue through the infant's first year of life.

Hospitalizations Patient hospitalization for diabetic control shall be recorded for data collection. Patients in the intervention group will not be contacted during their hospitalization. If medicine adjustments are made during their hospitalization, a reminder text message with the new regimen shall be sent the day after discharge. Contact will then resume by the above stated schedule. If a patient is hospitalized temporarily for a reason other than diabetes, contact will resume upon discharge. If the patient is hospitalized for the remainder of the pregnancy, the patient will be removed from the study. Triage visits will not be followed.

Delivery Delivery details will be abstracted from patient charts and shall include gestational age at delivery, fetal weight, vaginal versus cesarean delivery, incidence of shoulder dystocia, APGAR scores, and umbilical cord blood gases. The newborn chart shall be reviewed for the number of days spent in the neonatal intensive care unit, incidence of hypoglycemia and whether IV dextrose was required, and need for ventilator support or surfactant administration.

Maternal Complications Incidence of postpartum wound infections or dehiscence shall be collected.

Postpartum The postpartum glucose tolerance tests of women who had GDM will be reviewed to determine her glucose tolerance status.

Questionnaires/Surveys The participating patients will be asked to complete a survey upon entry into the study to identify barriers to their healthcare and their baseline knowledge of diabetes. A survey at the completion of their study (the postpartum visit or later) will be requested to evaluate patient perspectives on the study, their pregnancy and any perceived benefit from participation. The postpartum survey will be either completed at a postpartum visit, mailed to subjects, completed on line or subjects will be contacted by phone to complete the survey. If subjects do not return for a postpartum visit or do not complete the survey at that visit, three attempts will be made to contact subject for completion of the departure survey.

For participants who did not sign a version of the consent form that allowed for completion of the departure survey over the phone or online:

If their participation is ongoing, they will be approached at one of their visits and asked to review and sign an updated version of the consent form.

For subjects who have completed the pregnancy portion of their participation in the study but who did not complete a departure survey:

Subjects will be contacted over the phone to obtain permission to allow completion of this survey over the phone, by mail or online. A phone script will be used to contact patients. If subjects cannot be reached by phone, a letter will be sent to their home address. A maximum of three phone attempts will be made to contact subject.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is a pregnant person 18 years of age or older
2. The patient has been diagnosed with gestational diabetes or is a patient with known diabetes and a confirmed viable pregnancy
3. The pregnancy has a singleton pregnancy
4. The patient has access to a cellular phone with a text messaging plan

Exclusion Criteria:

1. The patient does not have a cellular phone
2. The patient becomes hospitalized for a pregnancy complication for the remainder of pregnancy
3. The fetus has a chromosomal or non-chromosomal malformation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
compliant diabetes care | up to 12 months
  Compliant with appointments, maintaining diabetes records, and medications, including glycemic control and pregnancy complications.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea Mostello, MD, Study Chair — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The data has been lost and we are in the process of trying to recover it.